CLINICAL TRIAL: NCT04709185
Title: Adrenal Venous Sampling Under 1 mg Overnight Dexamethasone Suppression Test to Determine Subtype in Primary Aldosteronism，a Single Center, Randomized, Double Blended, Placebo Controlled Clinical Trail
Brief Title: AVS After 1mg DST to Determine Subtype in PA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1mgDST AVS
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Primary Aldosteronism
Keywords: primary aldosteronism; adrenal venous sampling
MeSH Terms: conditions — Hyperaldosteronism | interventions — Dexamethasone; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVS after 1mg DST (Experimental): Patients divided into AVS after 1mg DST group need to oral 1mg dexamethasone the night before AVS
  Interventions: Drug: Dexamethasone 1 MG Oral Tablet
- AVS after placebo (Placebo Comparator): Patients divided into AVS after placebo group need to oral placebo the night before AVS
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone 1 MG Oral Tablet — oral 1 mg dexamethasone at 23:00-24:00 the night before AVS
  Arms: AVS after 1mg DST
Drug: Placebo — oral placebo at 23:00-24:00 the night before AVS
  Arms: AVS after placebo

SUMMARY:
To compare the effect of different procedures of AVS(after 1mg DST or not) in determining the subtypes and long-term outcomes of PA

DETAILED DESCRIPTION:
All paticipants will be randomly divided into 1mg DST group(Intervention group,n=43) and placebo group(Control group,n=43) and to determining the subtypes and to compare the long-term outcomes of patients with PA.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above, male or female, with legal capacity;
2. Patients who diagnosed as primary aldosteronism and willing to surgery

Exclusion Criteria:

1. Pregnant or lactating women
2. Patients with a history of malignant tumors or complicated with severe heart disease, eGFR<30ml/min/1.73m2, severe anemia (Hb<60g/L), stroke or acute coronary syndrome within 3 months, severe liver disease
3. Having contraindications or refusal to undergo AVS or unilateral adrenalectomy, or allergy to ACTH;
4. PA combined with Cushing syndrome (including subclinical Cushing); or considering glucocorticoid-suppressible aldosteronism (GRA) or adrenocortical carcinoma;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Complete biochemical remission | 1year
  Compare the rate of complete biochemical remission between two groups. Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.
Complete clinical remission | 1 year
  Compare the rate of complete clinical remission between two groups. Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.

SECONDARY OUTCOMES:
Daily defined doses of antihypertensive agents | 1 year
  The daily defined doses of antihypertensive agents of patients' blood pressure well controlled
Successful catheterization rate | procedure
  Calculate the successful rate of catheterization. Successful catheterization was defined as SI≥2 without ACTH stimulation or SI≥3 with ACTH stimulation.
Adverse events | 3 month
  Including adrenal venous hemorrhage and related adrenal insufficiency, hypertensive urgencies, anaphylactic shock, venous thrombosis, pulmonary embolism.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomu Li, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No